CLINICAL TRIAL: NCT05663450
Title: Extension of Resection After Positive Intraoperative Pathology During Surgery of Gastric and Gastroesophageal Junction Adenocarcinoma
Brief Title: Extended Resection After Positive Intraoperative Pathology in Gastric Cancer Surgery
Status: Completed | Type: Observational
Sponsor: University Hospital of Cologne (Other)
Responsible Party: Principal Investigator, Hakan Alakus, Clinical Professor and Senior Physician; Department of General, Visceral, Cancer and Transplantation Surgery, University Hospital of Cologne
Other Study IDs: HA_Pos_Margins_Gastrectomy
Record Dates: First submitted 2022-12-12; First posted 2022-12-23 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Gastric Cancer
Keywords: excision margin; prognosis; gastric cancer; resection
MeSH Terms: conditions — Stomach Neoplasms; Margins of Excision

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- patients with direct R0 (in primary intraoperative pathology consultation): patients undergoing (sub)total gastrectomy for gastric or GEJ adenocarcinoma with R0 without further resection (direct R0)
- patients with converted R0 (in second intraoperative pathology consultation): patients undergoing (sub)total gastrectomy for gastric or GEJ adenocarcinoma with R0 after positive IOC and extension of resection (converted R0)
- patients with remaining R1 (after final intraoperative pathology consultation): patients undergoing (sub)total gastrectomy for gastric or GEJ adenocarcinoma with R1 resection.

SUMMARY:
Of 737 consecutive patients undergoing (sub)total gastrectomy for gastric or GEJ adenocarcinoma, 679 cases with curative intent surgery between 05/1996 and 03/2019 were included. Patients were categorized into: i) R0 without further resection (direct R0), ii) R0 after positive IOC and extension of resection (converted R0) and iii) R1.

DETAILED DESCRIPTION:
This retrospective cohort study was performed at our tertiary referral center at the University Hospital of Cologne, Germany. Since 1st May 1996 medical charts of patients who undergo surgery for gastric or GEJ adenocarcinomas are collected in a department internal database for research analyses (Chairman since 05/2016 CJ Bruns, from 5/1996-4/2016 AH Hölscher).

In this study, patients undergoing curative surgery between 1st May 1996 and 31st March 2019 with (sub)total gastrectomy for gastric or GEJ adenocarcinoma were included. Palliative resections and resections with transthoracic esophagectomy and gastric pull-up were excluded.

Demographics, perioperative treatment, survival and clinicopathologic data were obtained. Medical records were reviewed and complications were categorized according to Clavien-Dindo classification.

Depending on IOCs, extended resection and final pathology report a treatment flow-chart was created (Figure 1): Patients were grouped on a) IOC received (yes/no), b) IOC positive (yes/no), c) extended resection (yes/no), d) second IOC (IOC2; yes/no), e) IOC2 positive (yes/no) and final pathology results (R0/R1). The decision to perform IOC and to carry out extended resection in case of positive IOC was at the discretion of the treating surgeon. Patients were then categorized into 3 subgroups according to final R status: R0 after extended resection (i.e. converted R0), R0 without extended resection (i.e. direct R0) and R1.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years
* tumor resection via total gastrectomy and subtotal esophagectomy

Exclusion Criteria:

* no additional other solid or hematological neoplasias in the medical history
* pregnancy
* surgical procedures in palliative intention

Ages: 59 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This retrospective cohort study was performed at our tertiary referral center at the University Hospital of Cologne, Germany. Since 1st May 1996 medical charts of patients who undergo surgery for gastric or GEJ adenocarcinomas are collected in a department internal database for research analyses (Chairman since 05/2016 CJ Bruns, from 5/1996-4/2016 AH Hölscher).
  In this study, patients undergoing curative surgery between 1st May 1996 and 31st March 2019 with (sub)total gastrectomy for gastric or GEJ adenocarcinoma were included.
Sampling Method: Non-Probability Sample
Enrollment: 679 (Actual)
Dates: Start 1996-05-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Rate of R1-resection during oncologic surgery | intraoperative pathology
  Rate of incomplete tumour resection (macroscopic: R2; microscopic: R1) during the surgical resection of gastric cancer patients

SECONDARY OUTCOMES:
Post-surgical survival | months (median follow-up: 29 months)
  post-surgical survival after radical surgical resection

CONTACTS AND LOCATIONS:
Overall Officials: Hakan Alakus, MD, Principal Investigator — University Hospital of Cologne

IPD SHARING:
Plan to Share IPD: Undecided
Data is available by the responsible PI on reasonable request

REFERENCES:
- [Derived] Plum PS, Barutcu AG, Pamuk A, Mallmann C, Chon SH, Chiapponi C, Dubbers M, Hellmich M, Moenig SP, Quaas A, Hoelscher AH, Bruns CJ, Alakus H. Extension of resection after positive intraoperative pathology during surgery for gastric and gastroesophageal junction adenocarcinoma: a retrospective cohort study. Int J Surg. 2023 Aug 1;109(8):2324-2333. doi: 10.1097/JS9.0000000000000484. PMID 37222663